CLINICAL TRIAL: NCT07034404
Title: Effects of a Digital Adapted Physical Activity Program on Physical Activity Levels and Sleep Quality in Patients With Spondyloarthritis: A Randomized, Controlled, Multicenter Study.
Brief Title: Effects of a Digital Exercise Intervention on Sleep and Physical Activity in Patients With Spondyloarthritis
Acronym: ASPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EssaiClinique_ASPIRE
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Spondylarthritis; Spondylarthropathies; Spondylitis, Ankylosing
Keywords: exercise; physical activity; sleep quality; digital intervention
MeSH Terms: conditions — Spondylarthritis; Spondylarthropathies; Spondylitis; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: Control (Standard treatment)
- Digital Adapted Physical Activity (Experimental)
  Interventions: Behavioral: Digital Adapted Physical Activity

INTERVENTIONS:
Behavioral: Digital Adapted Physical Activity — The digital Adapted Physical Activity (APA) program will be delivered via a digital platform and participants will be guided by an APA teacher to meet the WHO recommendations (i.e. 150 minutes of moderate intensity aerobic PA per week and muscle-strengthening activities that involve all major muscle groups twice weekly).
  Participants will benefit from 10 visits with the APA teacher: an initial assessment to define personalized goals and familiarize participants with the digital platform, eight sessions to monitor progress and adapt the exercise program, and a final evaluation aimed at assessing outcomes and encouraging long-term adherence to physical activity. Daily physical activity will be objectively monitored using a Withings connected watch to provide feedback and track metrics such as step count.
  Arms: Digital Adapted Physical Activity
Behavioral: Control (Standard treatment) — Participants will receive standard care and advice on physical activity (based on the recommendations of the World Health Organization, WHO, and the European Alliance of Associations for Rheumatology, EULAR) through a document provided to them.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess whether a tailored digital Adapted Physical Activity (APA) program can improve physical activity levels and sleep quality in adults diagnosed with spondyloarthritis (SpA).

The main questions it aims to answer are:

Does participation in a 6-month digital APA program increase average daily step count (measured with an activity tracker)? Does the program improve sleep quality (measured with the Pittsburgh Sleep Quality Index)? Researchers will compare participants receiving general physical activity advice (control group) to those following a structured digital APA program (intervention group) to see if the tailored digital support leads to better outcomes.

Participants will:

Complete baseline assessments including physical activity, sleep, pain, and quality of life measures.

Be randomly assigned to a control group or intervention group. For the intervention group, follow an individualized exercise program delivered through a virtual platform with support from an APA professional over 10 virtual sessions.

Wear a connected activity tracker (Withings) to monitor physical activity throughout the study.

Complete follow-up assessments at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80
* Followed in rheumatology for axial spondyloarthritis validating the ASAS or modified New York criteria at all stages of progression,
* Physically inactive (less than 150 minutes of moderate-intensity leisure-time physical activity per week), assessed at inclusion using the Global Physical Activity Questionnaire (GPAQ).
* With stable treatment for 3 months
* Signed informed consent
* Membership of a social security scheme
* Have access to a digital tool with an internet connection (tablet or smartphone)

Exclusion Criteria:

* Concurrent impairment by another osteoarticular pathology interfering with mobility of the spine or lower limbs,
* Central or peripheral neurological damage,
* Hip, knee or ankle arthroplasty performed or scheduled within 18 months,
* Any contraindication to physical activity (unstable or poorly controlled coronary ischaemia, severe asthma or significant obstructive ventilatory disorder (FEV1/FVC < 70%, FEV1 < 60% predicted), musculoskeletal pathology interfering with physical activity, proliferative retinopathy, macroscopic proteinuria, poorly controlled hypertension, etc.).
* Patients who do more than 150 minutes of moderate-intensity vigorous physical activity per week as part of their leisure activities.
* Persons covered by articles L1121-5 to L1121-8 of the Public Health Code
* Staff with a hierarchical link to the principal investigator

Non-inclusion criteria related to physical activity :

* Body mass index >35 kg/m2
* History of chest pain during physical activity
* History of sudden death in a first-degree relative
* History of thoracic irradiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Steps Per Day at 6 months | Baseline and 6 months
  Measured by Actigraph GT3X
Change from Baseline in Sleep Quality at 6 months | Baseline and 6 months
  Measured by the Pittsburgh Sleep Quality Index (PSQI) / A self-administered questionnaire / The 19 self-evaluation questions combine to yield 7 component scores, each scored from 0 to 3. A score of 0 indicates no difficulty, while a score of 3 indicates severe difficulty. The 7 component scores are summed to obtain a global score ranging from 0 (no difficulty) to 21 (major difficulties).

SECONDARY OUTCOMES:
Change in Steps Per Day from Baseline at 12 months | Baseline and 12 months
  Measured by Actigraph (GT3X)
Change in Sleep Quality from Baseline at 12 months | Baseline and 12 months
  Measured by the Pittsburgh Sleep Quality Index (PSQI) / A self-administered questionnaire / The 19 self-evaluation questions combine to yield 7 component scores, each scored from 0 to 3. A score of 0 indicates no difficulty, while a score of 3 indicates severe difficulty. The 7 component scores are summed to obtain a global score ranging from 0 (no difficulty) to 21 (major difficulties).
Change from Baseline in Total Sleep Time at 6 and 12 months | Baseline, 6 months and 12 months
  Measured using wrist-worn actigraphy (Actigraph GT3X)
Change from Baseline in Time Spent in Physical Activity at 6 and 12 months | Baseline, 6 months and 12 months
  Measured by time spent in light, moderate and sustained physical activity
Change from Baseline in Time Spent in Sedentary Behavior at 6 and 12 months | Baseline, 6 months and 12 months
  Measured by time spent awake in a seated or lying position measured by actimeter (Actigraph GT3X)
Change from Baseline in Sleep Quality at 6 and 12 months | Baseline, 6 months and 12 months
  Measured using wrist-worn actigraphy (Actigraph GT3X)
Change from Baseline in Fatigue at 6 and 12 months | Baseline, 6 months and 12 months
  Measured by the Pichot fatigue scale / Likert scale / This scale includes 8 items scored from 0 (strongly disagree) to 4 (strongly agree), with a total score ranging from 0 (no fatigue) to 32 (maximum fatigue)
Change from Baseline in Pain at 6 and 12 months | Baseline, 6 months and 12 months
  Measured by the visual analogue scale / Visual Analog Scale (VAS) / This scale consists of 1 item scored from 0 (no pain) to 10 (extreme pain)
Change from baseline in Disease Activity BASDAI to 6 and 12 months | Baseline, 6 months and 12 months
  Measured using questionnaires Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) / Self-administered scale / This scale consists of 6 items assessed on a numerical rating scale from 0 (not at all) to 10 (extremely). The overall score is the average of the six responses, giving a total score between 0 (no symptoms) and 10 (maximum symptoms).
Change from Baseline in Disease Activity ASDAS at 6 and 12 months | Baseline, 6 months and 12 months
  Measured using questionnaires Ankylosing Spondylitis Disease Activity Score (ASDAS) / A composite index combining several clinical variables and a biological marker of inflammation. The final score is calculated using a weighted formula, resulting in a continuous score / ASDAS values generally range from 0 to over 6, with the following thresholds:
  * < 1.3: Inactive disease
  * 1.3 to < 2.1: Moderate disease activity
  * 2.1 to < 3.5: High disease activity
  * ≥ 3.5: Very high disease activity
Change from Baseline in Functional Capacity at 6 and 12 months | Baseline, 6 months and 12 months
  Measured using questionnaires an Bath Ankylosing Spondylitis Functional Index (BASFI) / Self-administered questionnaire / This questionnaire consists of 10 items. Each item is scored on a numerical rating scale from 0 (no difficulty) to 10 (impossible). The final score is the average of the 10 responses, giving a total score between 0 (optimal functioning) and 10 (severely impaired functioning).
Change from Baseline in Quality of life ASAS-HI at 6 and 12 months | Baseline, 6 months and 12 months
  Measured using questionnaire ASAS-HI (Assessment of SpondyloArthritis International Society Health Index) / Likert-type scale / A questionnaire composed of 17 items. Each item is scored in a binary way (Agree = 1, Disagree = 0). The total score therefore ranges from 0 (best possible health) to 17 (significant health impairment).
Change from Baseline in Health-Related Quality of life at 6 and 12 months | Baseline, 6 months and 12 months
  Health-related quality of life (EQ-5D-5L) / 2 parts:
  * A descriptive system with 5 dimensions, each rated on 5 levels of severity (from 1 = no problems to 5 = extreme problems). The combination of responses defines a health state that can be converted into a single index value, generally ranging from -0.594 to 1, where 1 represents perfect health, 0 is equivalent to death, and negative values indicate a health state perceived as worse than death.
  * A visual analog scale ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change from Baseline in Cardiorespiratory fitness (VO2peak) at 6 months | Baseline, 6 months
  Cardiorespiratory stress test
Change from Baseline in Maximal Power Output at 6 months | Baseline, 6 months
  Maximal Power Output (watts)
Change from Baseline in Barriers and Facilitators to Physical Activity at 3, 6 and 12 months | Baseline, 3 months, 6 months and 12 months
  Measured using questionnaire Inflammatory Arthritis Facilitators and Barriers (IFAB) / A questionnaire consisting of 10 items / Elements that can be either barriers or facilitators are scored from -10 to 10. Items that are only barriers are scored from -10 to 0, and those that are only facilitators are scored from 0 to 10. When an item has no impact on physical activity, it is scored 0. If a question is missing, the item is scored 0. If two or more questions are missing, it is recommended not to compute the total score. The total score ranges from -70 to 70. Scores below -5 may justify targeted intervention.
Change from Baseline in Motivation for Physical Activity at 3, 6 and 12 months | Baseline, 3 months, 6 months and 12 months
  Measured using questionnaire motivational scale for physical activity for health purposes (EMAPS) / Questionnaire based on the self-determination theory / Composed of 18 items. Each item is scored on a 7-point Likert scale from 1 (does not correspond at all) to 7 (corresponds very strongly). Mean scores are calculated for each subscale / The questionnaire represents the following types of motivation:
  * Intrinsic motivation
  * Integrated motivation
  * Identified motivation
  * Introjected motivation
  * External motivation
  * Amotivation
Change from Baseline in Self-Esteem at 3, 6 and 12 months | Baseline, 3 months, 6 months and 12 months
  Measured using questionnaire Rosenberg scale / A self-assessment questionnaire composed of 10 items / Each item is rated on a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). The total score ranges from 10 to 40, with some items reverse-scored.
Change from Baseline in Pain Catastrophizing at 3, 6, 12 months | Baseline, 3, 6, 12 months
  Pain Castrophizing Scale / A self-administered questionnaire / It includes 13 items divided into 3 dimensions:
  * Rumination
  * Magnification
  * Helplessness / Each item is rated on a Likert scale from 0 (not at all) to 4 (all the time). The total score ranges from 0 to 52, with subscores for each dimension
Adherence to the Adapted Physical Activity Intervention | At 6 months
  Percentage of Physical Activity Sessions Completed by the Participant
Identify profiles of participants who are adherent or non- adherent to the Physical Activity Intervention according to personal determinants (motivation, beliefs) | At 6 months
  Adherent or non-adherent (adherence status defined as < 50% sessions completed)
Determine Sleep Quality Trajectories | Over 12 months
  Determine sleep quality trajectories based on data collected by the connected device (Sleel Analyzer, Withings) in the intervention group only
Intervention Satisfaction and Acceptability | At 6 months
  Perceived acceptability and satisfaction measured using a questionnaire in the intervention group

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Saint Etienne, Saint-Etienne